CLINICAL TRIAL: NCT07164677
Title: Efficacy of the Serratus Posterior Superior Intercostal Plane Block for Postoperative Acute Pain Management in Open-Heart Surgery
Brief Title: Serratus Posterior Superior Plane Block for Postoperative Pain in Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, BURHAN DOST, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPSIPB2025
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery; Post Operative Pain, Acute
Keywords: Cardiac surgery; Serratus Posterior Superior Plane Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A block randomization list will be created by a doctor who does not participate in patient follow-up using a web-based program, 'Research Randomizer (Urbaniak and Plous, 2013)'.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sealed opaque envelopes containing study participation numbers will be used to assign each patient. A researcher not involved in patient follow-up will use the web-based "Research Randomizer" (Urbaniak and Plous 2013) tool to give each participation number to a random group with a 1:1 ratio. A nurse not an active investigator in the study will have each participant choose an envelope containing the study participation number. They will inform the anesthetist administering the block/blocks about which group the patient is in immediately before administration. Researchers, surgeons, and nurses will not be aware of the randomization of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group SPSIP (Active Comparator): A bilaterally Serratus Posterior Superior Plane Block (60 ml, %0.25 bupivacaine, totally) + IV morphine patient-controlled analgesia (PCA)
  Interventions: Procedure: Bilateral ultrasound guided Serratus Posterior Superior Plane Block; Drug: IV morphine patient-controlled analgesia
- Group Control (Sham Comparator): A bilaterally Sham block + IV morphine patient-controlled analgesia (PCA)
  Interventions: Drug: IV morphine patient-controlled analgesia; Procedure: Bilateral ultrasound guided Sham Block

INTERVENTIONS:
Procedure: Bilateral ultrasound guided Serratus Posterior Superior Plane Block — Bilateral ultrasound-guided Serratus Posterior Superior Plane Block (total of 60 ml, %0.25 bupivacaine) will be performed Multimodal analgesia : Intraoperatively, all patients will receive 0.05 mg/kg (IBW) iv morphine. Thirty minutes before the end of surgery, 1 gram of intravenous paracetamol will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5mg/ml morphine. In cases where rescue analgesia is required (NRS score ≥4),iv fentanyl 25-50 mcg and/or ibuprofen and/or ketamine 10 mg will be administered. Patients are routinely administered iv dexamethasone 4 mg and IV 8 mg ondansetron 20 minutes before end of surgery for postoperative nausea and vomiting prophylaxis.
  Other Names: Serratus Posterior Superior Plane Block
  Arms: Group SPSIP
Drug: IV morphine patient-controlled analgesia — IV PCA of 0,5mg/ml morphine (the bolus dose is 20 μg/kg, the lock-in time of 6-10 minutes, the 4-hour limit is adjusted to be 80% of the calculated total amount).
  Other Names: morphine PCA
Procedure: Bilateral ultrasound guided Sham Block — Bilateral ultrasound-guided needle placement will be performed in the same anatomical plane as in the SPSIP group, but instead of local anesthetic, an equivalent volume of normal saline (30 mL per side) will be injected.
  Multimodal analgesia : Intraoperatively, all patients will receive 0.05 mg/kg (IBW) iv morphine. Thirty minutes before the end of surgery, 1 gram of intravenous paracetamol will be administered. Postoperative analgesia: iv paracetamol 1gr every 8 hours and IV PCA of 0,5mg/ml morphine. In cases where rescue analgesia is required (NRS score ≥4),iv fentanyl 25-50 mcg and/or ibuprofen and/or ketamine 10 mg will be administered. Patients are routinely administered iv dexamethasone 4 mg and IV 8 mg ondansetron 20 minutes before end of surgery for postoperative nausea and vomiting prophylaxis.
  Other Names: Sham Block
  Arms: Group Control

SUMMARY:
The aim of this study is to investigate the efficacy of bilateral serratus posterior superior intercostal plane (SPSIP) block on postoperative acute pain and opioid consumption in patients undergoing on-pump open-heart surgery. Postoperative outcomes including pain scores, cumulative morphine use, quality of recovery, and opioid-related side effects will be evaluated within the first 24 hours after surgery.

DETAILED DESCRIPTION:
Acute pain following cardiac surgery is a prevalent clinical problem that may negatively affect postoperative recovery, pulmonary function, and overall quality of life. Reported rates of moderate to severe pain after sternotomy range widely in the literature, largely due to factors such as vasospasm, heightened inflammatory responses, tissue and bone trauma during surgical dissection, and the placement of chest tubes. Although pain intensity usually subsides after the first 24 hours, inadequate analgesia during this critical period can prolong acute pain, delay mobilization, and increase the risk of chronic post-sternotomy pain syndrome.

Traditionally, neuraxial techniques such as thoracic epidural and paravertebral blocks have been used for pain management in cardiac surgery. However, their application remains controversial due to technical difficulties and patient-related risks, including coagulation disorders, complete heparinization, hemodynamic instability, and potential complications such as pneumothorax. In recent years, fascial plane chest wall blocks, including serratus anterior, parasternal blocks and erector spinae plane blocks, have gained traction as safer alternatives, particularly in patients receiving antiplatelet or anticoagulant therapy.

The serratus posterior superior intercostal plane (SPSIP) block, first described in 2023, represents a novel approach for thoracic analgesia, providing extensive dermatomal coverage from C3 to T10. By targeting the fascial plane between the serratus posterior superior and intercostal muscles, this block offers the potential for effective analgesia across cervical and thoracic regions. Preliminary reports and case series have demonstrated its promising role in thoracic and minimally invasive cardiac surgery.

This prospective, randomized, double-blind, parallel-group trial will evaluate the efficacy of bilateral SPSIP block in patients undergoing on-pump open-heart surgery. Participants will be allocated to either:

SPSIP Group: General anesthesia + SPSIP Block + Patient-Controlled Analgesia (PCA)

Control Group: General anesthesia + Sham Block + PCA

The primary outcome is cumulative morphine consumption during the first 24 postoperative hours. Secondary outcomes include acute pain scores at rest and with movement, time to first opioid demand, rescue analgesia requirements, incidence of postoperative nausea and vomiting (PONV), opioid-related side effects, intraoperative remifentanil consumption, and quality of recovery assessed by the QoR-15 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 undergoing elective on-pump open-heart surgery via median sternotomy.
* American Society of Anesthesiologists (ASA) classification II-III patients.
* Patients who can use PCA.
* Patients who will sign the informed consent form.

Exclusion Criteria:

* History of opioid use for more than four weeks
* Chronic pain syndromes
* Patients with a history of local anesthetic or opioid allergy, hypersensitivity
* Alcohol and drug addiction
* Conditions where regional anesthesia is contraindicated
* Failure in the dermatomal examination performed after the block
* Emergency surgeries and redo surgeries.
* Individuals with obstructive sleep apnea.
* Left ventricular ejection fraction less than 30%.
* Patients with severe psychiatric illnesses (such as psychosis, dementia) that limit cooperation with verbal numerical pain scales.
* Pregnant and breastfeeding patients.
* Hematological disorders.
* Significant impairment in the function of a major organ (e.g., severe hepatic or renal disease). • Patients who cannot be extubated within the first 6 hours postoperatively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption in the first 24 hours after surgery | Postoperative day 1
  The primary outcome will be defined as cumulative opioid consumption during the first 24 hours following surgery, which will be calculated in intravenous morphine milligram equivalents (IV-MME), encompassing both PCA- administered morphine and rescue intravenous tramadol, according to the standardized ESAIC conversion guidelines. Patients can request opioids via a PCA device when their NRS score is≥ 4.

SECONDARY OUTCOMES:
Cumulative opioid consumption in the first 12 hours after surgery | Postoperative12 hours
  The secondary outcome will be defined as cumulative opioid consumption during the first 12 hours following surgery, calculated in intravenous morphine milligram equivalents (IV-MME). This will include both PCA-administered morphine and rescue intravenous tramadol, in accordance with the standardized ESAIC conversion guidelines. Patients may request opioids using a PCA device when their NRS score is ≥ 4.
Numerical Rating Scale Assessment of Postoperative Pain | Postoperative day 1
  Pain scores will be assessed using the 11-point Numerical Rating Scale (NRS), where 0 indicates no pain and 10 represents the worst imaginable pain. Evaluations will be performed both at rest (static) and during coughing or deep breathing (dynamic). Assessments will be conducted in the post-anesthesia care unit (PACU) after extubation and once communication is established, and subsequently at 3, 6, 12, 18, and 24 hours postoperatively.
Intraoperative Remifentanil Consumption | The remifentanil consumption will be recorded from anesthesia induction until the patient is referred to the recovery unit, up to 250 minutes
  Total intraoperative remifentanil consumption will be recorded in micrograms (μg) from the start of anesthesia induction until the end of surgery.
Time to First Opioid Demand via PCA | Postoperative day 1
  Defined as the time elapsed from the patient's arrival in the post-anesthesia care unit (PACU) to the first patient- initiated opioid request via the patient-controlled analgesia (PCA) device.
The number of patients who required rescue analgesia. | Postoperative day 1
  he number of patients who required additional IV tramadol due to breakthrough pain (NRS ≥4) despite PCA use.
The patient number of Rescue antiemetic Requirement | Postoperative day 1
  All patients received standard prophylaxis for postoperative nausea and vomiting (PONV), including 8 mg IV dexamethasone before induction and 0.15 mg/kg IV ondansetron (based on ideal body weight) approximately 20 minutes before the end of surgery. PONV was assessed at 0, 3, 6, 12, 18, and 24 hours after extubation using a 5- point scale (0 = no nausea to 4 = multiple episodes of vomiting). Patients with a PONV score ≥3 received rescue treatment with 10 mg IV metoclopramide in 100 mL normal saline via slow infusion. The number of patients requiring rescue antiemetic therapy was recorded.
The number of patients with complications | Postoperative 7 days on an average
  The number of patients has any complications -directly related to the block or the drug used in the block- will be recorded
Patients' satisfaction and quality of pain management | preoperative day 1 and Postoperative day 1
  Patients' pain management satisfaction and quality will be evaluated using the QoR-15 score. The QoR-15 consists of 5 test areas: pain (2 questions), physical comfort (5 questions), physical state (2 questions), psychological state (2 questions), and emotional state (4 questions). Each question is rated on a 10-point scale ranging from 0 = "never" to 10 = "always" (scoring is reversed for negative questions). QoR-15 Turkish Version will be used for assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Burhan Dost, Study Director — Ondokuz Mayis University, Samsun, Atakum 55139
Locations (1):
- Burhan Dost, Samsun, Turkey (Türkiye)